CLINICAL TRIAL: NCT02816658
Title: The Role of the Robotic Platform in Inguinal Hernia Repair Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Michael Rosen, Director, Cleveland Clinic Comprehensive Hernia Center, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-1594
Record Dates: First submitted 2016-05-26; First posted 2016-06-28 (Estimated); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic Surgery (Active Comparator): Laparoscopic Inguinal Hernia Repair through a Transabdominal, Preperitoneal Approach
  Interventions: Other: Laparoscopic Inguinal Hernia Repair
- Robotic Surgery (Active Comparator): Robotic Inguinal Hernia Repair
  Interventions: Other: Robotic Inguinal Hernia Repair

INTERVENTIONS:
Other: Laparoscopic Inguinal Hernia Repair — Laparoscopic Inguinal Hernia Repair
  Arms: Laparoscopic Surgery
Other: Robotic Inguinal Hernia Repair — Robotic Inguinal Hernia Repair
  Arms: Robotic Surgery

SUMMARY:
Inguinal hernia repair is one of the most commonly performed general surgery operations. However, to date, the ideal surgical approach for inguinal hernia surgery. The investigators therefore, propose a randomized controlled trial comparing laparoscopic inguinal hernia surgery repair to robotic inguinal hernia repair surgery.

The investigators hypothesize that the robotic approach to inguinal hernia repair will result in improved post-operative outcomes compared to traditional laparoscopic inguinal hernia repairs.

Specific Aim #1: To determine if the robotic approach will result in a significant reduction in postoperative pain and earlier return to full function when compared to a laparoscopic inguinal hernia repair.

Specific Aim #2: To perform a cost analysis to determine the financial implications of performing a robotic versus a laparoscopic inguinal hernia repair.

Specific Aim #3: To determine the effect of surgeon reported ergonomics when performing laparoscopic versus robotic inguinal hernia repairs.

Specific Aim #4: Evaluate the long term hernia recurrence rates associated with laparoscopic versus robotic inguinal hernia repairs.

DETAILED DESCRIPTION:
Inguinal hernia repair is the most commonly performed general surgery procedure in the United States. Despite the prevalence of this procedure, there is no consensus regarding the optimal approach to this surgical procedure. Since the advent of the laparoscopic inguinal hernia repair in 1990, there is a growing body of research that has investigated the efficacy of this minimally invasive surgical approach. To date, the laparoscopic approach to inguinal hernia repair has proven beneficial in reducing post-operative pain and allowing for earlier return to normal activity versus the traditional open inguinal hernia repair. In addition, the laparoscopic approach to inguinal hernia repair has been advocated for recurrent inguinal hernia repairs and bilateral inguinal hernia repairs.

Despite these advantages, however, there are several limitations of the laparoscopic inguinal hernia repair. Specifically, unstable camera platforms, two-dimensional imaging, rigid laparoscopic instruments, and poor surgeon ergonomics make the laparoscopic approach to inguinal hernia repair challenging. Furthermore, the learning curve associated with a laparoscopic inguinal hernia repair has been prohibitive for many surgeons. Finally, the laparoscopic approach to inguinal hernia repair often requires the utilization of some form of fixation device, such as surgical tacks, which have been associated with chronic pain, vascular injury, as well as increased overall cost of the operation. The robotic platform has been shown to help compensate for many of these short-comings of laparoscopic surgery as it provides three-dimensional imaging, improved instrument mobility, articulation, suturing capability (which allows for a more cost-effective procedure with decreased risk of post-operative chronic pain), and surgeon comfort. Because of these reasons, it is important to determine the specific advantages the robotic approach will provide for inguinal hernia repairs.

The laparoscopic approach to inguinal hernia repair has proven beneficial in reducing post-operative pain and earlier returns to normal activity versus the traditional open inguinal hernia repair. However, the overall penetrance of laparoscopic inguinal hernia repair has remained consistently below 20% of all inguinal hernia procedures performed in the United States. The robotic platform provides several potential advantages over the laparoscopic inguinal hernia repair including three dimensional visualization, the ability to suture (rather than tack) the mesh, as well as the ability to suture the peritoneal defect closed. This technological platform could provide earlier adoption and proficiency for surgeons to perform a minimally invasive inguinal hernia repair with improved surgical outcomes. As more general surgeons begin to incorporate robotic surgery into their practice, the robotic platform might provide further improvements in the outcomes of minimally invasive inguinal hernia repair over even traditional laparoscopic inguinal hernia repair.

The investigators propose a Randomized Clinical Trial comparing the robotic versus laparoscopic inguinal hernia repair techniques. The investigators hypothesize that the robotic approach to inguinal hernia repair will result in improved post-operative outcomes compared to traditional laparoscopic inguinal hernia repairs.

Specific Aim #1: To determine if the robotic approach will result in a significant reduction in postoperative pain and earlier return to full function when compared to a laparoscopic inguinal hernia repair.

Specific Aim #2: To perform a cost analysis to determine the financial implications of performing a robotic versus a laparoscopic inguinal hernia repair.

Specific Aim #3: To determine the effect of surgeon reported ergonomics when performing laparoscopic versus robotic inguinal hernia repairs.

Specific Aim #4: Evaluate the long term hernia recurrence rates associated with laparoscopic versus robotic inguinal hernia repairs.

ELIGIBILITY:
Inclusion Criteria:

1. 21 years or older
2. No prior open abdominal surgery at or below the umbilicus
3. Primary or recurrent unilateral inguinal hernia repair
4. No previous preperitoneal mesh placement
5. BMI less than or equal to 40kg/m2

Exclusion Criteria:

1. Need for an open inguinal hernia repair
2. Patients presenting for evaluation of bilateral inguinal hernias
3. Patients requiring surgical repair of a strangulated inguinal hernia
4. Patients with liver disease defined by the presence of ascites
5. Patients with end-stage renal disease requiring dialysis
6. Patients who are unable to give informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-05; Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Pain Score | 2 Years
  Differences in postoperative pain between those patients who undergo robotic inguinal hernia repair versus laparoscopic inguinal hernia repair.

SECONDARY OUTCOMES:
Ergonomic Tool | 2 Years
  Differences in surgeon ergonomics between the two approaches as measured by the NASA-TLX and RULA ergonomic assessments.
Institution cost analysis | 2 Years
  Total cost of the operation for the two approaches.
Long-term recurrence rate differences | 2 Years
  Comparison of recurrence rates, as assessed by an independed, blinded assessor

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Rosen, MD, Principal Investigator — The Cleveland Clinic
Locations (6):
- United States (6):
  - Washington University, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Greenville Health System, Greenville, South Carolina
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prabhu AS, Carbonell A, Hope W, Warren J, Higgins R, Jacob B, Blatnik J, Haskins I, Alkhatib H, Tastaldi L, Fafaj A, Tu C, Rosen MJ. Robotic Inguinal vs Transabdominal Laparoscopic Inguinal Hernia Repair: The RIVAL Randomized Clinical Trial. JAMA Surg. 2020 May 1;155(5):380-387. doi: 10.1001/jamasurg.2020.0034. PMID 32186683